CLINICAL TRIAL: NCT02946970
Title: Brain Responses to Intragastric Administration of a Bitter Agonist in Homeostatic and Hedonic Brain Regions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S57915
Record Dates: First submitted 2016-05-12; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
MeSH Terms: interventions — Quinine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Intragastric infusion
  Interventions: Other: Control
- Quinine hydrochloride (Experimental): Intragastric infusion
  Interventions: Other: Quinine hydrochloride

INTERVENTIONS:
Other: Quinine hydrochloride — Intragastric administration of a bitter tastant agonist (10 μmol/kg quinine-hydrochloride)
  Arms: Quinine hydrochloride
Other: Control — Intragastric administration of distilled water
  Arms: Control

SUMMARY:
The investigators aim to study the brain mechanisms underlying the effect of subliminal (not consciously perceived) intragastric administration of bitter tastants on hunger and food intake, which was previously found. The investigators will assess brain activation patterns after an acute intragastric administration of Quinine-hydrochloride versus saline on two different test days, and will simultaneously assess a putative role of altered gut peptide release in these effects. The hypothesis is that intragastric infusion of a bitter agonist will decrease the activity in homeostatic and hedonic brain regions and that this effect is mediated by gut peptide release.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Female
* N = 15
* Age 18 - 60
* Body Mass Index (BMI) of 20 - 25 kg/m
* Stable body weight for at least 3 months prior to the start of the study

Exclusion Criteria:

* Abdominal or thoracic surgery. Exception: appendectomy
* Gastrointestinal, endocrine or neurological diseases
* Cardiovascular, respiratory, renal or urinary diseases
* Hypertension
* Food or drug allergies
* Anemia
* Eating disorders and people who show abnormal eating behavior
* Depressive disorders
* Psychotic disorders
* No medication on a regular basis, expect for oral contraception
* Conditions that can interfere with functional magnetic resonance imaging (fMRI), e.g. cochlear implants, metal fragments or metal implants in the body, pacemaker, neural stimulator, …
* No history of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Alcohol abuse (more than 21 units of alcohol for men, more than 14 units for woman per week)
* Dieters
* Pregnant or breastfeeding women
* Claustrophobia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Functional brain images | From the start of the study until 50 minutes after the start of the study
  Change in brain responses after administration compared to baseline will be assessed via functional magnetic resonance imaging.

SECONDARY OUTCOMES:
hunger scores | every 10 minutes since the scan starts until until 50 minutes after the start of the scan
  The hunger scores will be taken every 10 minutes since the scan starts via a 10 cm visual analogue scale.
Ghrelin levels | every 10 min since the scan starts until 50 minutes after the start of the scan.
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure ghrelin levels by radioimmuno-assay.
Motilin levels | every 10 min since the scan starts until 50 minutes after the start of the scan
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure motilin levels by radioimmuno-assay.
CCK levels | every 10 min since the scan starts until 50 minutes after the start of the scan
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure CCK levels by radioimmuno-assay.
PYY levels | every 10 min since the scan starts until 50 minutes after the start of the scan
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure PYY levels by Enzyme-Linked Immuno Sorbent Assay
GLP-1 levels | every 10 min since the scan starts until 50 minutes after the start of the scan
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure GLP-1 levels by Enzyme-Linked Immuno Sorbent Assay

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof, Principal Investigator — University of Leuven

IPD SHARING:
Plan to Share IPD: No